CLINICAL TRIAL: NCT05554133
Title: Precision Optical Guidance for Oral Biopsy Based on Next-Generation Hallmarks of Cancer (1R01DE029590-01): A Clinical Study to Evaluate and Optimize the Technical Performance Characteristics of an Active Biopsy Guidance System
Brief Title: Precision Optical Guidance for Oral Biopsy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2020-1115; NCI-2022-07929 (Other: NCI-CTRP Clinical Trials Registry); R01DE029590-01 (NIH)
Record Dates: First submitted 2022-09-20; First posted 2022-09-26 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Oral Lesions
MeSH Terms: interventions — Proflavine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- The Active Biopsy Guidance System (Experimental): This imaging scanning device is made up of 2 parts: the optical mapping scope and the high-resolution microendoscope (HRME):
  Interventions: Device: High Resolution Microendoscope (HRME); Device: Optical Mapping Scope; Drug: Proflavine hemisulfate

INTERVENTIONS:
Device: High Resolution Microendoscope (HRME) — The High Resolution Microendoscope (HRME) take pictures of a very small area of the lining of the mouth, about the size of a pencil tip, but at high magnification.
Device: Optical Mapping Scope — The optical mapping scope displays a wide area of the lining of the mouth (about the size of the top of a soda can) by shining different colors of light into the mouth and taking pictures.
Drug: Proflavine hemisulfate — A coloring substance (a fluorescent dye which glows green in the dark), called proflavine hemisulfate, will be painted on areas of the mouth with a cotton tip applicator to help improve the pictures

SUMMARY:
To learn if a new type of imaging device called the Active Biopsy Guidance System can help doctors to decide when and where to perform invasive biopsies of mouth lesions.

DETAILED DESCRIPTION:
Primary objective:

-To evaluate and optimize the technical performance characteristics of an Active Biopsy Guidance System.

Secondary objective:

-To provide a preliminary estimate of the sensitivity and specificity of the Active Biopsy Guidance System with respect to histopathology. Optical imaging; optical projection of light onto tissue; optical contrast agent (proflavine).

ELIGIBILITY:
Inclusion Criteria:

1. Adult subjects with clinically evident oral lesions such as leukoplakia or erythroplakia, oral potentially malignant disorders (OPMD) such as lichen planus and graft vs. host disease, pathologic diagnosis of dysplasia, squamous cell carcinoma, or a history of resected oral cancer, are eligible to participate. Patients with previous treatment including surgery, radiation, chemotherapy or other therapies are also eligible.
2. Ability to understand and willingness to sign a written Informed Consent Document (ICD).

Exclusion Criteria:

1. Known allergy to proflavine or acriflavine.
2. Age less than 18 years.
3. Pregnant or nursing females.
4. Adults unable to consent
5. Prisoners and other vulnerable populations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-06-15 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
To establish a preliminary estimate of the sensitivity and specificity of the Active Biopsy Guidance System with respect to histopathology | Through study completion an average of 1 year.

CONTACTS AND LOCATIONS:
Overall Officials: Ann Gillenwater, MD, Principal Investigator — MD Anderson Caner Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org